CLINICAL TRIAL: NCT04500665
Title: Anti-Inflammatory Treatment of Uremic Cardiomyopathy With Colchicine
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Leo F. Buckley, PharmD, Clinical Pharmacy Specialist, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020P002468; K23HL150311 (NIH)
Record Dates: First submitted 2020-07-30; First posted 2020-08-05 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Colchicine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Colchicine (Experimental): Colchicine 0.3 mg once daily
  Interventions: Drug: Colchicine
- Placebo (Placebo Comparator): Placebo once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Colchicine — Colchicine
  Arms: Colchicine
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study is designed to determine the efficacy and safety of colchicine in patients with chronic kidney disease.

ELIGIBILITY:
A. Inclusion Criteria:

* Age 21 years to 80 years (inclusive)
* eGFR of 15 to 75 mL/min per 1.73 m2
* Urine albumin-to-creatinine ratio of greater than 30 mg/g
* Use of maximally tolerated doses of an angiotensin-converting enzyme inhibitor or angiotensin receptor blocker if urine albumin-to-creatinine ratio greater than 300 mg-g
* Use of a sodium-glucose co-transporter-2 inhibitor if indicated in the opinion of the participant's primary clinician
* Willing and able to provide written informed consent and to adhere to the study protocol

B. Exclusion Criteria:

1. History of intolerance or allergy to colchicine
2. Hospitalization for any reason within the previous 30 days
3. Acute condition that requires emergent treatment in the opinion of a physician investigator
4. Stage C or D heart failure according to ACC-AHA criteria77
5. Left ventricular ejection fraction less than 40%
6. Symptomatic valvular heart disease
7. Congenital heart disease (corrected or uncorrected)
8. History of orthotopic heart transplant
9. Kidney failure, defined as kidney transplant recipient or requirement for hemodialysis or peritoneal dialysis
10. Worsening kidney function or acute kidney injury, defined as an increase in serum creatinine of greater than 0.3 mg/dL in the previous 30 days or 50% within the previous 7 days
11. Use of immunosuppressive or anti-inflammatory medications within the previous 30 days, with the exception of less than 5 days of non-steroidal anti-inflammatory drugs or corticosteroids for acute pain or other acute conditions that have since fully resolved provided that the last dose of non-steroid anti-inflammatory drug was at least 7 days before enrollment
12. Familial Mediterranean Fever, gout (unless no flare within the previous 12 months), pericarditis or other indications for colchicine treatment
13. Use of systemic antimicrobial therapy within the previous 30 days or active infection
14. History of respiratory illness that, in the opinion of a physician investigator, may increase the risk of pneumonia
15. Surgery within the previous 30 days or surgery planned to occur within the expected study period
16. Current malignancy or receipt of treatment for malignancy within the previous 1 year
17. Frailty or life-expectancy shortened by comorbidity such as cancer that would increase the participant's risk in the opinion of a physician investigator
18. Neutrophil count < 2,000 cells/mm3
19. Platelet count < 50,000 cells/mm3
20. Concomitant use of a P-gp inhibitor (e.g., cyclosporine, ranolazine, digoxin) and/or moderate-strong CYP3A4 inhibitor (e.g., clarithromycin, indinavir, itraconazole, ritonavir, nefazodone, diltiazem, verapamil, grapefruit juice, fluconazole)
21. Medications that may cause myopathy or rhabdomyolysis (i.e., simvastatin, gemfibrozil, fenofibrate) , a creatine kinase level after the run-in period that exceeds the upper limit of the normal laboratory reference range (if baseline was below the upper limit) or that increases by 50% or more from pre- to post-run-in
22. Moderate-severe hepatic disease (Child-Pugh B or C)
23. Pregnant or unwilling/unable to assure appropriate contraception
24. Breastfeeding

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-11-11 (Estimated)

PRIMARY OUTCOMES:
Between-group change in left ventricular global longitudinal strain | 4 weeks
  Assessed using transthoracic echocardiography

SECONDARY OUTCOMES:
Between-group change in left ventricular systolic and diastolic function | 4 weeks
  Assessed using transthoracic echocardiography
Between-group change in left ventricular volumes | 4 weeks
  Assessed using transthoracic echocardiography
Between-group change in left ventricular size | 4 weeks
  Assessed using transthoracic echocardiography
Between-group change in systemic inflammation | 4 weeks
  Assessed using C-reactive protein

CONTACTS AND LOCATIONS:
Overall Officials: Leo F Buckley, PharmD MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No